CLINICAL TRIAL: NCT05569122
Title: The Utility of pGz in Primary Mitochondrial Disorders
Brief Title: Applying pGz in Mitochondrial Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-018532
Record Dates: First submitted 2022-07-07; First posted 2022-10-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Mitochondrial Myopathies; Mitochondrial Diseases
Keywords: Passive Exercise; periodic acceleration
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Aim 1 will have the 3 study interventions/study visits occur in random order. The interventions will be performed in primary mitochondrial disease patients and healthy controls
  Aim 2 will have all participants complete the study interventions/visits in the same order. Patients will be from the PICU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aim 1: Primary Mitochondrial Disease Patients (Experimental): The participant has the interventions/study visits occur in a random order:
  CPET pGz administration through pGz Bed pGz administration through Gentle Jogger
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing; Device: pGz Bed; Device: Gentle Jogger; Drug: Lumason® contrast agent
- Aim 1: Healthy Controls (Experimental): The participant has the interventions/study visits occur in a random order:
  pGz administration through Gentle Jogger CPET pGz administration through pGz Bed
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing; Device: pGz Bed; Device: Gentle Jogger; Drug: Lumason® contrast agent
- Aim 2: PICU Patients (Experimental): All participants in Aim 2 will have the interventions/study visits occur in the same order: Exercise Pedal and Gentle Jogger
  Interventions: Device: Gentle Jogger; Device: Exercise Pedal; Drug: Lumason® contrast agent

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Testing — Testing with an exercise bicycle that is considered "standard of care" for determination of exercise capacity. Participants will complete about 20 minutes of pedaling in a stationary exercise bike
  Arms: Aim 1: Healthy Controls; Aim 1: Primary Mitochondrial Disease Patients
Device: pGz Bed — Participants will lay down on a passive exercise (pGz) bed for 45 minutes during which the bed will administer passive exercise through periodic acceleration
  Arms: Aim 1: Healthy Controls; Aim 1: Primary Mitochondrial Disease Patients
Device: Gentle Jogger — Participants will have passive exercise delivered through the gentle jogger device for 45 minutes. This may be sitting down (aim 1 participants) or laying down (aim 2 participants)
Device: Exercise Pedal — Participants will exercise while laying down for 20 minutes with an exercise pedal that attaches to the bed
  Arms: Aim 2: PICU Patients
Drug: Lumason® contrast agent — Contrast agent used during a vascular ultrasound of the upper leg. Will occur at each study visit twice before and after pGz bed, gentle jogger, exercise pedal or CPET. Drug Administration will be through an IV line and take about 5 - 10 minutes.

SUMMARY:
This is a multi-aim study, studying the effects of conventional exercise (measured through Cardiopulomary Exercises Testing or an in-bed pedal exercise) and passive exercise through periodic acceleration (pGz). Aim 1 will focus on the differences between primary mitochondrial disease (PMD) patients and healthy volunteers. Aim 2 is an exploratory aim, which will be studying the effects in patients admitted to the Children's Hospital of Philadelphia Pediatric Intensive Care Unit (PICU).

DETAILED DESCRIPTION:
Aim 1: Primary Mitochondrial Disease Patients and Healthy Controls

Individuals will be screened for eligibility for study entry, and answer questions relating to their ability to perform study procedures and their physical activity levels. Individuals who meet study criteria will have 3 study visits, and each study visit will involve a different intervention.

At each of these study visits, individuals will complete one of the following interventions: Cardiopulmonary Exercise Testing (CPET), pGz administration through a bed or recliner, and pGz through a device called a Gentle Jogger. While participants will complete all three study visits, the order of the study visits will occur in random order.

During the study visits, participants will have blood draws before and after the study intervention, a vascular ultrasound with a Lumason contrast agent before and after the study intervention, and a Creatine Chemical Exchange Saturation Transfer (CrCEST) MRI of the lower leg.

Aim 2: Patients in the Pediatric Intensive Care Unit (PICU)

Individuals will be screened for eligibility for study entry. Individuals who meet study criteria will have 2 study visits during their admission to the PICU. The first study visit will involve a pedal exercise and the second study visit will involve pGz administration through a device called a Gentle Jogger.

During the study visits, participants will have blood draws before and after the study intervention, a vascular ultrasound with a Lumason contrast agent before and after the study intervention, and if able to safely complete, an CrCEST MRI of the lower leg.

ELIGIBILITY:
Aim 1 Enrollment Criteria Inclusion Criteria for Healthy Controls

* Males or females, 10 years to 60 years, with a minimum height for participation of 135 cm
* Ambulatory and able to complete routine clinical exercise testing
* Willing and able to complete all study procedures
* For individuals under the age of 18, parental/guardian permission (informed consent) and as appropriate, child assent
* For individuals over the age of 18 the ability to provide informed consent

Inclusion Criteria for PMD Patients

* Males or females, 10 years to 60 years, with a minimum height for participation of 135 cm
* Ambulatory and able to complete routine clinical exercise testing
* Willing and able to complete all study procedures
* Genetically confirmed mitochondrial myopathy (MM) as defined by a diagnosis of primary mitochondrial disease (PMD) with predominant symptoms of myopathy as expressed by exercise intolerance and muscle weakness and fatigue
* Parental/guardian permission (informed consent) and as appropriate, child assent

Exclusion Criteria for All Aim 1 Participants General Exclusion Criteria

* Tracheostomy
* Non-ambulatory
* Unable to complete routine exercise testing
* Diagnosed with or have symptoms of vertigo
* Within 1 month of a recent hospital admission for acute illness
* Severe co-existing cardiac or pulmonary disease
* Cognitive impairment that may preclude ability to comply with study procedures
* Pregnant or lactating females
* Active alcohol and/or substance abuse
* At the discretion of the principal investigator (PI), any medical condition that will interfere with or prevent the safe completion of the study
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures
* Use of investigational agent(s) within 4 weeks
* Individuals who are employed by the U.S. Department of Defense, including U.S military personal
* Patients with biliary atresia with asplenia or polysplenia.
* Patients with prior liver transplant.
* Patients with cystic fibrosis.
* Patients with chronic lung disease.
* Patients with portal vein thrombosis, cavernous transformation of the portal vein or absent portal vein.
* Patients with significant heart disease or severe congenital heart disease.
* Patients with a history of allergic reaction to Lumason®, sulfur hexafluoride, sulfur hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol, distearoylphosphatidlycholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na, palmitic acid) or other components of the ultrasound contrast agent
* Any history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic evaluation
* Any history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation
* Past or current employment involving (or exposure to) a metal grinder (e.g., at a construction worksite)
* Claustrophobia or any known medical conditions which can be exacerbated by stress, anxiety, or panic attacks triggered by enclosed spaces
* Inability to lie flat in an MRI scanner for up to 45 minutes
* Unable to perform sub-maximal ankle dorsiflexion leg exercise during the MRI study

Aim 2 Enrollment Criteria Inclusion Criteria for PICU PMD Non-Ambulatory Patients

* Males or females ages 10 to 23 years (children and adults)
* Non-ambulatory
* Genetically confirmed mtDNA-PMD
* Cooperative and capable of following research procedures
* Have cognitive ability to enable cooperation with study procedures
* Admitted to the PICU with an anticipated length of stay for >24 hours
* Willing and able to complete all study procedures
* For individuals under the age of 18, parental/guardian permission (informed consent) and as appropriate, child assent
* For individuals over the age of 18 the ability to provide informed consent

Inclusion Criteria for PICU non-PMD neuromuscular diagnosis

* Males or females ages 10 to 23 years (children and adults)
* Non-ambulatory
* Genetically confirmed non-PMD neuromuscular diagnosis
* Cooperative and capable of following research procedures
* Have cognitive ability to enable cooperation with study procedures
* Admitted to the PICU with an anticipated length of stay for >24 hours
* For individuals under the age of 18, parental/guardian permission (informed consent) and as appropriate, child assent
* For individuals over the age of 18 the ability to provide informed consent

Inclusion Criteria for all other PICU Participants

* Males or females ages 10 to 23 years (children and adults)
* Non-ambulatory
* No known genetic diagnosis with healthy pre-morbid status, admitted to PICU
* Cooperative and capable of following research procedures
* Have cognitive ability to enable cooperation with study procedures
* Admitted to the PICU with an anticipated length of stay for >24 hours
* Willing and able to complete all study procedures
* For individuals under the age of 18, parental/guardian permission (informed consent) and as appropriate, child assent
* For individuals over the age of 18 the ability to provide informed consent

Exclusion Criteria for All Aim 2 Participants

* Have cognitive impairment that may preclude ability to comply with study procedures
* Have cardiorespiratory instability
* Patients in whom are so sick that they will not be able to cooperate with the study procedures
* Have clear contraindications to mobilization
* Have fixed lower limb deformities/contractures that would prohibit lower extremity exercise
* Pregnant or lactating females
* Active alcohol and/or substance abuse
* At the discretion of the principal investigator (PI), any medical condition that will interfere with or prevent the safe completion of the study
* Use of investigational agent(s) within 4 weeks
* Individual who are employed by the U.S. Department of Defense, including U.S military personal
* Patients with biliary atresia with asplenia or polysplenia.
* Patients with prior liver transplant.
* Patients with cystic fibrosis.
* Patients with chronic lung disease.
* Patients with portal vein thrombosis, cavernous transformation of the portal vein or absent portal vein.
* Patients with significant heart disease or severe congenital heart disease.
* Patients with a history of allergic reaction to Lumason®, sulfur hexafluoride, sulfur hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol, distearoylphosphatidlycholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na, palmitic acid) or other components of the ultrasound contrast agent

Exclusion Criteria Specific to study procedure: CrCEST MRI Scan:

* Any history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic evaluation
* Any history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation
* Past or current employment involving (or exposure to) a metal grinder (e.g., at a construction worksite)
* Claustrophobia or any known medical conditions which can be exacerbated by stress, anxiety, or panic attacks triggered by enclosed spaces
* Inability to lie flat in an MRI scanner for up to 45 minutes
* Unable to perform sub-maximal ankle dorsiflexion leg exercise during the MRI study

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Mean Difference in Maximal Oxygen Consumption between primary mitochondrial disease patients and healthy volunteers | During Cardiopulmonary Exercise Testing, which will last 1 hour
  Maximal Oxygen Consumption will be measured only during CPET
Aim 2: Arterial-Venous (A-V) O2 difference | A total of 4 15 minute blood draws
  This will be measured through blood draws that occur before and after study interventions
Aim 1 and 2: Oxygen Consumption | 1 hour per study intervention
  Measured During the study interventions

SECONDARY OUTCOMES:
Aim 1 and 2: A/B ratio measurement through EKG or Plethsymography | 1 hour per study intervention
  To measure hemodynamic physiologic marker of cardiac output (CO)
Aim 1 and 2: Heart Rate | 1 hour per study intervention
  To measure hemodynamic physiologic marker of cardiac output (CO)
Aim 1 and 2: OXPHOS Capacity | Aim 1 subjects will complete 2 1 hour MRIs, Aim 2 Subjects will complete 1 1-hour MRI
  Measured through a CrCEST Leg MRI, which measures creative levels and recovery in the leg
Aim 1 and 2: Plasma Lactate Levels | 15 minute blood draws that occur pre and and immediately after each study intervention
  Measured through venous blood draws
Aim 1 and 2: Vasodilatation | 30 minute ultrasound that occurs pre and immediately after each study intervention
  Measured through a vascular ultrasound with contrast
NO release | 15 minutes, before and immediately after each study intervention
  Measured through Plethsymography
Plasma Nom Levels | 15 minute blood draws that occur pre and immediately after each study intervention
  Measured through venous blood draws
Post-operative Patient Satisfaction Survey | 15 minutes, taken after each study intervention
  Participant tolerance to pGz compared to CPET
Borg Scale | 15 minutes, taken after each study intervention
  Participant tolerance to pGz compared to CPET

CONTACTS AND LOCATIONS:
Overall Officials: Zuela Zolkipli-Cunningham, MBChB, MRCP, Principal Investigator — Attending Physician
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Sackner MA, Lopez JR, Banderas V, Adams JA. Can Physical Activity While Sedentary Produce Health Benefits? A Single-Arm Randomized Trial. Sports Med Open. 2020 Oct 2;6(1):47. doi: 10.1186/s40798-020-00278-3. PMID 33006749
- [Background] Sackner MA, Patel S, Adams JA. Changes of blood pressure following initiation of physical inactivity and after external addition of pulses to circulation. Eur J Appl Physiol. 2019 Jan;119(1):201-211. doi: 10.1007/s00421-018-4016-7. Epub 2018 Oct 22. PMID 30350153
- [Background] Burstein DS, McBride MG, Min J, Paridon AA, Perelman S, Huffman EM, O'Malley S, Del Grosso J, Groepenhoff H, Paridon SM, Brothers JA. Normative Values for Cardiopulmonary Exercise Stress Testing Using Ramp Cycle Ergometry in Children and Adolescents. J Pediatr. 2021 Feb;229:61-69.e5. doi: 10.1016/j.jpeds.2020.09.018. Epub 2020 Sep 11. PMID 32926876
- [Background] Taivassalo T, Jensen TD, Kennaway N, DiMauro S, Vissing J, Haller RG. The spectrum of exercise tolerance in mitochondrial myopathies: a study of 40 patients. Brain. 2003 Feb;126(Pt 2):413-23. doi: 10.1093/brain/awg028. PMID 12538407
- [Background] Tarnopolsky M. Exercise testing in metabolic myopathies. Phys Med Rehabil Clin N Am. 2012 Feb;23(1):173-86, xii. doi: 10.1016/j.pmr.2011.11.011. Epub 2011 Dec 11. PMID 22239882
- [Background] Tarnopolsky M. Exercise testing as a diagnostic entity in mitochondrial myopathies. Mitochondrion. 2004 Sep;4(5-6):529-42. doi: 10.1016/j.mito.2004.07.011. Epub 2004 Sep 30. PMID 16120411
- [Background] Taivassalo T, Haller RG. Exercise and training in mitochondrial myopathies. Med Sci Sports Exerc. 2005 Dec;37(12):2094-101. doi: 10.1249/01.mss.0000177446.97671.2a. PMID 16331135
- [Background] Adams JA, Uryash A, Bassuk J, Sackner MA, Kurlansky P. Biological basis of neuroprotection and neurotherapeutic effects of Whole Body Periodic Acceleration (pGz). Med Hypotheses. 2014 Jun;82(6):681-7. doi: 10.1016/j.mehy.2014.02.031. Epub 2014 Mar 12. PMID 24661939
- [Background] Adams JA, Mangino MJ, Bassuk J, Kurlansky P, Sackner MA. Regional blood flow during periodic acceleration. Crit Care Med. 2001 Oct;29(10):1983-8. doi: 10.1097/00003246-200110000-00022. PMID 11588467
- [Background] M. Fujita et al., "Periodic acceleration enhances release of nitric oxide in healthy adults," Int. J. Angiol., vol. 14, no. 1, pp. 11-14, Feb. 2005, doi: 10.1007/s00547-005-2013-2.
- [Background] Uryash A, Bassuk J, Kurlansky P, Altamirano F, Lopez JR, Adams JA. Antioxidant Properties of Whole Body Periodic Acceleration (pGz). PLoS One. 2015 Jul 2;10(7):e0131392. doi: 10.1371/journal.pone.0131392. eCollection 2015. PMID 26133377
- [Background] Uryash A, Bassuk J, Kurlansky P, Altamirano F, Lopez JR, Adams JA. Non-invasive technology that improves cardiac function after experimental myocardial infarction: Whole Body Periodic Acceleration (pGz). PLoS One. 2015 Mar 25;10(3):e0121069. doi: 10.1371/journal.pone.0121069. eCollection 2015. PMID 25807532
- [Background] Adams JA, Patel S, Lopez JR, Sackner MA. The Effects of Passive Simulated Jogging on Short-Term Heart Rate Variability in a Heterogeneous Group of Human Subjects. J Sports Med (Hindawi Publ Corp). 2018 Oct 1;2018:4340925. doi: 10.1155/2018/4340925. eCollection 2018. PMID 30402499
- [Background] Sackner MA, Gummels E, Adams JA. Nitric oxide is released into circulation with whole-body, periodic acceleration. Chest. 2005 Jan;127(1):30-9. doi: 10.1378/chest.127.1.30. PMID 15653959
- [Background] Adams JA, Bassuk J, Wu D, Grana M, Kurlansky P, Sackner MA. Periodic acceleration: effects on vasoactive, fibrinolytic, and coagulation factors. J Appl Physiol (1985). 2005 Mar;98(3):1083-90. doi: 10.1152/japplphysiol.00662.2004. Epub 2004 Oct 22. PMID 15501928
- [Background] Betik AC, Parker L, Kaur G, Wadley GD, Keske MA. Whole-Body Vibration Stimulates Microvascular Blood Flow in Skeletal Muscle. Med Sci Sports Exerc. 2021 Feb 1;53(2):375-383. doi: 10.1249/MSS.0000000000002463. PMID 32826637
- [Background] Sjoberg KA, Rattigan S, Hiscock N, Richter EA, Kiens B. A new method to study changes in microvascular blood volume in muscle and adipose tissue: real-time imaging in humans and rat. Am J Physiol Heart Circ Physiol. 2011 Aug;301(2):H450-8. doi: 10.1152/ajpheart.01174.2010. Epub 2011 May 27. PMID 21622816
- [Background] Kogan F, Haris M, Debrosse C, Singh A, Nanga RP, Cai K, Hariharan H, Reddy R. In vivo chemical exchange saturation transfer imaging of creatine (CrCEST) in skeletal muscle at 3T. J Magn Reson Imaging. 2014 Sep;40(3):596-602. doi: 10.1002/jmri.24412. Epub 2013 Oct 31. PMID 24925857
- [Background] DeBrosse C, Nanga RPR, Wilson N, D'Aquilla K, Elliott M, Hariharan H, Yan F, Wade K, Nguyen S, Worsley D, Parris-Skeete C, McCormick E, Xiao R, Cunningham ZZ, Fishbein L, Nathanson KL, Lynch DR, Stallings VA, Yudkoff M, Falk MJ, Reddy R, McCormack SE. Muscle oxidative phosphorylation quantitation using creatine chemical exchange saturation transfer (CrCEST) MRI in mitochondrial disorders. JCI Insight. 2016 Nov 3;1(18):e88207. doi: 10.1172/jci.insight.88207. PMID 27812541
- [Background] Jeppesen TD, Schwartz M, Olsen DB, Wibrand F, Krag T, Duno M, Hauerslev S, Vissing J. Aerobic training is safe and improves exercise capacity in patients with mitochondrial myopathy. Brain. 2006 Dec;129(Pt 12):3402-12. doi: 10.1093/brain/awl149. Epub 2006 Jun 30. PMID 16815877